CLINICAL TRIAL: NCT00006461
Title: Systemic Chemotherapy, Second Look Surgery and Conformal Radiation Therapy Limited to the Posterior Fossa and Primary Site for Children >/= to 8 Months and <3 Years With Non-metastatic Medulloblastoma: A Children&Apos;s Oncology Group Phase III Study
Brief Title: Combination Chemotherapy Followed by Second-Look Surgery and Radiation Therapy in Treating Children With Nonmetastatic Medulloblastoma or Primitive Neuroectodermal Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P9934; NCI-2012-02362 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068269 (Other: Clinical Trials.gov); POG-P9934 (Other: Pediatric Oncology Group); COG-P9934 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Untreated Childhood Medulloblastoma; Untreated Childhood Supratentorial Primitive Neuroectodermal Tumor
MeSH Terms: interventions — Cisplatin; Cyclophosphamide; Vincristine; Etoposide; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy, surgery, radiation therapy (Other): Patients receive induction chemotherapy consisting of vincristine sulfate IV on days 1, 8, and 15; cisplatin IV over 6 hours on day 1; cyclophosphamide IV over 30 minutes on day 2; and oral etoposide daily on days 2-22. Treatment repeats every 28 days for a total of 4 courses. After completion of induction chemotherapy, patients with residual disease undergo a therapeutic conventional surgery (second resection). Within 4 weeks after completion of induction chemotherapy or second resection, patients receive 3-dimensional conformal radiation therapy daily, 5 days a week, for 6 weeks. Four weeks after completion of 3-dimensional conformal radiation therapy, patients receive alternating treatments of maintenance chemotherapy. Patients receive vincristine sulfate IV on days 1, 8, and 15 and cyclophosphamide IV over 30 minutes on day 1 of courses 1, 3, 5, and 7 and oral etoposide daily on days 1-21 of courses 2, 4, 6, and 8. Treatment continues every 28 days for 8 courses.
  Interventions: Drug: cisplatin; Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: etoposide; Procedure: therapeutic conventional surgery; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: etoposide — Given PO
  Other Names: EPEG; VP-16; VP-16-213
Procedure: therapeutic conventional surgery — Undergo surgery
Radiation: 3-dimensional conformal radiation therapy — Undergo 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT

SUMMARY:
This phase III trial is studying how well combination chemotherapy followed by second-look surgery and radiation therapy works in treating children with nonmetastatic medulloblastoma or primitive neuroectodermal tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and combining chemotherapy with surgery and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the proposed treatment for children >= 8.0 months and < 3 years of age at registration with non-metastatic (M0) medulloblastoma is more effective than the combined treatments given to children of the same age and extent of disease on POG 9233, as measured by event-free survival (EFS) rates.

SECONDARY OBJECTIVES:

I. To assess the feasibility and safety of the planned use of second look surgery and focal conformal radiation therapy following chemotherapy. II. To determine the acute and chronic toxicities associated with the above treatment regimens.

III. To describe the neuropsychological and neuroendocrine effects of this systemic chemotherapy, surgery, and local, conformal radiation. IV. To determine the feasibility and validity of a centralized telephone interview based data collection method for neuropsychological evaluations. V. To determine the incidence of atypical teratoid/rhabdoid tumor (AT/RT) in children enrolled on this study.

OUTLINE: This is a multicenter study.

Patients receive induction chemotherapy consisting of vincristine IV on days 1, 8, and 15; cisplatin IV over 6 hours on day 1; cyclophosphamide IV over 30 minutes on day 2; and oral etoposide daily on days 2-22. Treatment repeats every 28 days for a total of 4 courses. After completion of induction chemotherapy, patients with residual disease undergo a second resection. Within 4 weeks after completion of induction chemotherapy or second resection, patients receive focal conformal radiotherapy daily, 5 days a week, for 6 weeks. Four weeks after completion of radiotherapy, patients receive alternating treatments of maintenance chemotherapy. Patients receive vincristine IV on days 1, 8, and 15 and cyclophosphamide IV over 30 minutes on day 1 of courses 1, 3, 5, and 7 and oral etoposide daily on days 1-21 of courses 2, 4, 6, and 8. Treatment continues every 28 days for 8 courses. Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary medulloblastoma or posterior fossa primitive neuroectodermal tumor

  * Prior definitive tumor resection within 6 weeks of study
* No evidence of metastases
* Hemoglobin at least 10 g/dL
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* AST less than 2.5 times normal
* Bilirubin less than 1.5 mg/dL
* Creatinine less than 1.2 mg/dL
* Creatinine clearance greater than 70 mL/min
* No prior chemotherapy
* No prior radiotherapy
* See Disease Characteristics

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2000-10; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Event-free survival rate | 1 year

SECONDARY OUTCOMES:
Acute and chronic toxicities associated with the treatment regimens | Up to 9 years
Neuropsychological and neuroendocrine effects of this systemic chemotherapy, surgery, and local, conformal radiation | Up to 9 years
Feasibility and validity of a centralized telephone interview based data collection method for neuropsychological evaluations | Up to 9 years
Incidence of atypical teratoid and/or rhabdoid tumor | Up to 9 years

CONTACTS AND LOCATIONS:
Overall Officials: David Ashley, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States